CLINICAL TRIAL: NCT05578547
Title: Effect of Combined Kendell and McKenzie Postural Correction Exercises on Brachial Plexus Mechanosensitivity in Chronic Non-Specific Neck Pain
Brief Title: Effect of Combined Kendell and McKenzie on Brachial Plexus Mechanosensitivity in Chronic Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, lecturer of physical therapy Basic Science department faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT.012/003920
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Chronic Non-Specific Neck Pain
Keywords: Kendell Postural Correction Exercises; McKenzie Postural Correction Exercises; Brachial Plexus Mechanosensitivity; Chronic Non-Specific Neck Pain
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined Kndell and McKenzie group (Experimental): patients receivee combined Kndell and McKenzie cervical posture correction exercises, ultrasound, hot packs, cervical extensors stretching and strengthening exercise.
  Interventions: Other: combined Kendell and McKenzie cervical posture correction exercises, ultrasound, hot packs, cervical extensors stretching and strengthening exercise.
- Conventional therapy group (Active Comparator): patients receive ultrasound, hot packs, cervical extensors stretching and strengthening exercise.
  Interventions: Other: ultrasound, hot packs, cervical extensors stretching and strengthening exercise.

INTERVENTIONS:
Other: combined Kendell and McKenzie cervical posture correction exercises, ultrasound, hot packs, cervical extensors stretching and strengthening exercise. — • The combined exercise will be done as follow:
  1) slowly pull the subject's neck to the head, thereby attaching the chin to the neck.
  (2) the subject's eyes should be looking directly forward. (3) hold both hands on the back of the subject's head. (4) ask the subject to push his/her head backwards against the hands. (5) ask for the hands to be spread as wide as possible in order to stretch the pectoralis major.
  Therapeutic ultrasound:
  Moist heat packs:
  Stretching Exercises:
  Posture correction exercises training for forward head posture includes stretching of tight muscles such as Pectoralis major, levator scapulae, upper trapezius, suboccipital muscles, sternocleidomastoid Stretching exercises of pectoralis major, levator scapulae, upper fibres of trapezius, suboccipital muscles, sternocleidomastoid Strengthening Exercises Chin Tucks exercise Neck isometric exercises
  Arms: combined Kndell and McKenzie group
Other: ultrasound, hot packs, cervical extensors stretching and strengthening exercise. — Therapeutic ultrasound:
  Moist heat packs:
  Stretching Exercises:
  Posture correction exercises training for forward head posture includes stretching of tight muscles such as Pectoralis major, levator scapulae, upper trapezius, suboccipital muscles, sternocleidomastoid Stretching exercises of pectoralis major, levator scapulae, upper fibres of trapezius, suboccipital muscles, sternocleidomastoid Strengthening Exercises Chin Tucks exercise Neck isometric exercises
  Arms: Conventional therapy group

SUMMARY:
this study will apply a modified cervical exercise that combined McKenzie's and Kendall's exercises, consisted of neck extension exercises and stretching of the pectoralis muscles at the same time. Although they only required a short time to complete, the exercises proved being effective in improving forward head posture.

DETAILED DESCRIPTION:
Nowadays, neck pain is predictable among people of all ages, whether it is a golden-ager, juvenile, or a schoolchild. In any stage of life, a person may experience neck pain because of the poor posture and prolonged use of electronic devices. Students spend about 80% of their daily life in college and performing various activities in their college, like slouching over computers and laptops for long periods for their college projects, backpacks over one shoulder (laptop bag), and squeezing into chairs or desk, etc. All are posture ruining activities that every student perform daily

When there is no traumatic injury, poor posture is the main root of neck pain. Bad posture results with the functional deviation from the normal aligned posture without any structural changes in the spine or lower extremities (Saxton, 1993). In reflection, muscle weakness and muscular imbalance of the musculoskeletal system leads to the postural deformities that coincide with muscle findings. Continuous load on the neck leads to disc collapse or degenerative changes in the future.

Several studies reported the effect of cervical postural correction exercises on pain, ROM and cranio-cervical angle in patients with chronic non-specific neck pain. Few studies have been concerned with measuring mechanosensitivity as an indicator technique of the effect of different modalities on chronic non-specific neck pain. With the proposal of the combined Kendall and McKenzie exercise program for patients with chronic non-specific neck pain secondary to forward head posture deviations recently, it is important to document how could this new combined technique impact neck posture as well as neural tissue sensitivity and function.

The outcome of this study will provide necessary information to clarify the effect of combined Kendall and McKenzie exercise program on mechanosensitivity and peripheral nerve excitability, pain intensity and cervical range of motion. This study may help and add to the physiotherapists exercise protocol for patient with chronic non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty subjects of both genders will be recruited in the study.
2. The age of the recruited subjects will be ranging from 25 to 50 years old
3. Subjects having neck pain symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature, for at least the last 3 months )
4. Subjects with a craniovertebral angle (CVA) of less than 54º
5. Subjects with a BMI between 25-30 )

Exclusion Criteria:

1. History of previous injury of the neck
2. History of surgical intervention at the neck
3. History of inflammatory joint disease affecting facet joints
4. Neurological disorders such as cervical spondylosis, spondylolythesis or disc prolapse
5. Rheumatic diseases.
6. Cancer patients.
7. Patients who received pain medication or physical therapy for their neck pain during the last 3 months
8. Patients who are unable to perform the exercises.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Neck pain intensity will be measured with a visual analogue scale (VAS) | at first week and after 4 weeks of treatment
Change in Cervical ROM will be measured by CROM | at first week and after 4 weeks of treatment
The strength-duration curve to assess the change in mechanosensitivity of brachial plexus | at first week and after 4 weeks of treatment
Change in Functional performance will be measured by Neck disability index | at first week and after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university, Giza, Egypt